CLINICAL TRIAL: NCT06197555
Title: Comparision of the Clinical Efficacy of Different Desensitizing Toothpastes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Sevdenur GÜNENÇ, Dentist, Altinbas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/138
Record Dates: First submitted 2023-12-12; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Dentine Hypersensitivity
Keywords: Dentin Hypersensitivity; Toothpaste; Fluoride; Arginine; Nano-Hydroxyapatite
MeSH Terms: conditions — Dentin Sensitivity | interventions — fluorophosphate; Tin Fluorides; nano-hydroxyapatite-collagen; Arginine; Calcium Carbonate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Sodium Monofluorophosphate) (Active Comparator): Dentifrice containing Sodium Monofluorophosphate, daily homecare usage Colgate®, Cavity Protection
  Interventions: Other: Sodium Monofluorophosphate
- Group B (Stannous Fluoride) (Active Comparator): Dentifrice containing Stannous Fluoride, daily homecare usage Oral B®, Gum Calm & Sensitivity
  Interventions: Other: Stannous Fluoride
- Group C (Nano-Hydroxyapatite) (Active Comparator): Dentifrice containing Nano-Hydroxyapatite, daily homecare usage ApaCare®
  Interventions: Other: Nano-Hydroxyapatite
- Group D (8% Arginine & Calcium Carbonate) (Active Comparator): Dentifrice containing 8% Arginine & Calcium Carbonate, daily homecare usage Colgate®, Sensitive Pro-Relief
  Interventions: Other: 8% Arginine & Calcium Carbonate

INTERVENTIONS:
Other: Sodium Monofluorophosphate — Test toothpaste, participants will brush selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least one minute. The method of application of these agents will be the fingertip method. Patients continued to use the paste twice daily, morning and evening, for 16 weeks.
  Arms: Group A (Sodium Monofluorophosphate)
Other: Stannous Fluoride — Test toothpaste, participants will brush selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least one minute. The method of application of these agents will be the fingertip method. Patients continued to use the paste twice daily, morning and evening, for 16 weeks.
  Arms: Group B (Stannous Fluoride)
Other: Nano-Hydroxyapatite — Test toothpaste, participants will brush selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least one minute. The method of application of these agents will be the fingertip method. Patients continued to use the paste twice daily, morning and evening, for 16 weeks.
  Arms: Group C (Nano-Hydroxyapatite)
Other: 8% Arginine & Calcium Carbonate — Test toothpaste, participants will brush selected sensitive teeth each for 30 seconds followed by the whole mouth thoroughly for at least one minute. The method of application of these agents will be the fingertip method. Patients continued to use the paste twice daily, morning and evening, for 16 weeks.
  Arms: Group D (8% Arginine & Calcium Carbonate)

SUMMARY:
Dentin hypersensitivity is a common problem in society. Untreated hypersensitivity affects the patient's quality of life, complicates plaque control and increases the risk of caries and periodontal disease. This study aimed to evaluate the clinical efficacy of desensitizing toothpastes containing sodium fluoride, stannous fluoride, nano-hydroxyapatite, 8% arginine and calcium carbonate.

Fourty eight patients with at least two teeth with positive responses to air and mechanical stimulus were included in the study and were divided into four groups. Sodium fluoride (Colgate®, Cavity Protection) in group A, stannous fluoride (Oral B® Gum Calm & Sensitivity) in group B, nano-hydroxyapatite (ApaCare®) in group C and 8% arginine and calcium carbonate combination in group D (Colgate® Sensitive Pro- ReliefTM) were used by the patients continuously for 16 weeks. Dentin hypersensitivity, by using VAS and Shiff scores and periodontal parameters were evaluated at baseline, 2nd week, 4th week and last 16th week.

ELIGIBILITY:
Inclusion Criteria:

* Dentin hypersensitivity complaints
* Systemically healthy
* Not during pregnancy & lactation
* No sensitivity treatment in the last 6 months
* Forty-eight patients with positive response to VAS and Schiff tests were included.

Exclusion Criteria:

People who have;

* Any systemic disease
* Take regular medication for any other reason
* Undergone periodontal surgery within the last 6 months,
* History of allergy to toothpaste materials,
* Active caries, restoration and/or bridge on the sensitive tooth,
* Orthodontic appliances,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity Reduction | Baseline, 2nd week, 4th week, 16th week
  Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Hypersensitivity Reduction | Baseline, 2nd week, 4th week, 16th week
  The Schiff Scale examiner covers the adjacent teeth on either side of the patient's hypersensitive tooth with his/her fingers. Air from the tip of the dental unit's air-water sprayer is applied to the cervical region of the hypersensitive tooth at a distance of approximately 1 cm for 1 second. The degree of hypersensitivity is scored according to the Schiff cold air sensitivity scale. Scoring :
  Score 0: The individual does not respond to the stimulus. Score 1: The individual responds to the stimulus but does not request its termination. Score 2: The individual responds to the stimulus and requests its termination or moves to avoid the stimulus. Score 3: The individual responds to the stimulus, finds the stimulus painful and requests its termination. The pain persists for a few seconds after the stimulus is terminated.

SECONDARY OUTCOMES:
Clinical Periodontal Measurements | Baseline, 16th week
  Probing depths (mm)
Clinical Periodontal Measurements | Baseline, 16th week
  Clinical attachment levels (mm)
Clinical Periodontal Measurements | Baseline, 16th week
  Plaque score (%),
Clinical Periodontal Measurements | Baseline, 16th week
  Bleeding score (%)

CONTACTS AND LOCATIONS:
Overall Officials: İlknur ÖZENCİ, Study Chair — Altinbas University; Şebnem DİRİKAN İPÇİ, Study Director — Altinbas University; Gökser ÇAKAR, Study Director — Altinbas University; Sevdenur GÜNENÇ, Principal Investigator — Altinbas University
Locations (1):
- Altinbas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided